CLINICAL TRIAL: NCT03369067
Title: Real-Time Monitoring and Glucose Control During Winter-Sport Exercise in Youth With Type 1 Diabetes: The AP Ski Camp Continued
Brief Title: Artificial Pancreas and Remote Monitoring During a T1DM Youth Ski Camp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Tandem Diabetes Care, Inc. (Industry); DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Marc Breton, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20335
Record Dates: First submitted 2017-11-15; First posted 2017-12-11 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Artificial Pancreas (AP); Continuous Glucose Monitor (CGM); Closed Loop Control (CLC); Insulin Pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Pancreas, Artificial; Continuous Glucose Monitoring; Insulin Infusion Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Artificial Pancreas Therapy (Experimental): Subjects will use the Tandem t:slim X2 with Control-IQ Technology + Dexcom G6 to automatically modulate their insulin delivery and control their glycemia. In addition a Dexcom G5 Share/Follow system will be used to remote monitor the participants and ensure safety.
  Interventions: Device: Tandem t:slim X2 with Control-IQ Technology + Dexcom G6; Device: Dexcom CGM G5
- Sensor Augmented Pump Therapy (Placebo Comparator): Subjects will use a Dexcom CGM G5 and their Continuous Subcutaneous Insulin Infusion devices (insulin pumps) to modulate their insulin delivery and control their glycemia. In addition a Dexcom G5 Share/Follow system will be used to remote monitor the participants and ensure safety.
  Interventions: Device: Dexcom CGM G5; Device: Continuous Subcutaneous Insulin Infusion

INTERVENTIONS:
Device: Tandem t:slim X2 with Control-IQ Technology + Dexcom G6 — Subjects will use the Tandem t:slim X2 with Control-IQ Technology and Dexcom G6 CGM to control their glycemia. The Tandem t:slim X2 with Control-IQ device is an automated insulin delivery pump that automatically adjusts insulin delivery to predicted and prevailing glucose levels, as measured by a Dexcom G6 continuous glucose monitor [CGM].
  Other Names: Artificial Pancreas; Automated Insulin Delivery Device
  Arms: Artificial Pancreas Therapy
Device: Dexcom CGM G5 — The Dexcom G5 CGM is a subcutaneous glucose sensor that provides an estimate of the prevailing blood glucose concentration approximately every 5 minutes.The Dexcom G5 sensor alerts the user if the prevailing glucose concentration is higher or lower than predetermined thresholds, or if it is changing too fast. In addition, the Share/Follow functionality of the Dexcom G5 allows up to 5 people ("followers") to receive in real-time information about the current blood glucose concentration and rate of change.
  The Dexcom G5 system will be used by participants and clinical study staff to monitor glucose levels 24h/day during the camp, ensure participants safety, and compute glycemic control outcomes
  Other Names: Continuous Glucose monitoring
Device: Continuous Subcutaneous Insulin Infusion — Subjects will use a subcutaneous pump to deliver insulin and control their glycemia.
  Other Names: Insulin pump
  Arms: Sensor Augmented Pump Therapy

SUMMARY:
An early feasibility study that will test the efficacy of the Tandem t:slim X2 with Control-IQ and Dexcom Continuous Glucose System G6 in a winter/ski camp environment.

DETAILED DESCRIPTION:
This proposal aims to demonstrate the superiority of the Closed-Loop Control (CLC), also known as Artificial Pancreas (AP) named Tandem t:slim X2 with Control-IQ Technology and assess usability in a supervised setting in a controlled environment compared with state-of-the-art Sensor-Augmented Pump (SAP) therapy for the treatment of type 1 diabetes (T1D) in adolescents. Phase 1 participants (13-18 years old) and Phase 2 participants (6-12 years old) will be assessed during a ~48 hour ski camp; Upon completion of the ski camp, Phase 2 participants (6-12 years old) will also be assessed during a ~78 hour home use.

ELIGIBILITY:
Inclusion Criteria:

1. Criteria for documented hyperglycemia (at least 1 must be met):

   * Clinical diagnosis of type 1 diabetes (C-peptide levels and antibody determinations are not required)
   * The diagnosis of type 1 diabetes is based on the investigator's judgment
2. Criteria for requiring insulin at diagnosis (both criteria must be met):

   * Daily insulin therapy for ≥ 6 months
   * Insulin pump therapy for ≥ 3 months (note: must be willing to disable any glucose suspend, predictive suspend, or artificial pancreas functionality on insulin pump during study)
3. Virginia camp: age 13-18 years; Colorado/Stanford camps: 6-12 years
4. Avoidance of acetaminophen-containing medications (i.e. Tylenol) while wearing the continuous glucose monitor.
5. Willingness to wear a continuous glucose sensor and physiological monitor for the duration of the study
6. Not being pregnant at the start of the trial. All female subjects of childbearing potential will be screened for pregnancy.

8. If the participant is less than 13 years of age and the parents or the study team request it, at least one parent commit to stay with the study subject at the camp site 9. A parent/caregiver is available for system training and will commit to be the main responsible person for the use of the AP system at home

Exclusion Criteria:

1. Diabetic ketoacidosis in the past 6 months
2. Hypoglycemic seizure or loss of consciousness in the past 6 months
3. History of seizure disorder (except for hypoglycemic seizure)
4. History of any heart disease including coronary artery disease, heart failure, or arrhythmias
5. History of altitude sickness
6. Chronic pulmonary conditions that could impair oxygenation
7. Cystic fibrosis
8. Current use of oral glucocorticoids, beta-blockers or other medications, which in the judgment of the investigator would be a contraindication to participation in the study.
9. History of ongoing renal disease (other than microalbuminuria).
10. Subjects requiring intermediate or long-acting insulin (such as NPH, Detemir or Glargine).
11. Subjects requiring other anti-diabetic medications other than insulin (oral or injectable).
12. Pregnancy
13. Presence of a febrile illness within 24 hours of start ski camp or acetaminophen use while wearing the CGM. The camp study subject will not participate in the trial if these conditions are met.
14. Medical or psychiatric condition that in the judgment of the investigator might interfere with the completion of the protocol such as (for parent and/or child):

    * Inpatient psychiatric treatment in the past 6 months
    * Uncontrolled adrenal insufficiency
    * Alcohol abuse

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Breton, PhD, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (3):
- United States (3):
  - Stanford University, Stanford, California
  - Barbara Davis Center, University of Colorado, Aurora, Colorado
  - University of Virginia Center for Diabetes Technology, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Result] Ekhlaspour L, Forlenza GP, Chernavvsky D, Maahs DM, Wadwa RP, Deboer MD, Messer LH, Town M, Pinnata J, Kruse G, Kovatchev BP, Buckingham BA, Breton MD. Closed loop control in adolescents and children during winter sports: Use of the Tandem Control-IQ AP system. Pediatr Diabetes. 2019 Sep;20(6):759-768. doi: 10.1111/pedi.12867. Epub 2019 May 23. PMID 31099946

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization occurred at the ski camp after check In. Forty-eight were randomized, participated, and completed the study (24 in UVA, 12 in Colorado, and 12 at Stanford).
Groups:
- Experimental AP Group: The experimental AP Group used the Tandem t:slim X2 with Control-IQ Technology (Tandem Diabetes Care, San Diego, CA) which was integrated with the Dexcom G6 CGM (Dexcom, San Diego, CA).
- Control SAP Group: The control SAP group used their home insulin pumps. All participants were fitted with a Dexcom CGM G5 continuous glucose monitor with Share™ capability with minimum calibration before breakfast and dinner (7:00 A.M. and 7:00 P.M.) using a study-provided blood glucose meter (BGM) (ContourNext Link; Ascencia Diabetes Care, Parsippany, NJ).
Period: Overall Study
Arm/Group | Experimental AP Group | Control SAP Group
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental AP Group | Control SAP Group | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 48 participated and completed the study (24 in UVA, 12 in Colorado, and 12 at Stanford). One subject signed consent but didn't met eligibility (no history of pump use), and five subjects left the study after a change in the Stanford camp dates (blizzard cancellation).
  years
    Stanford: number analyzed (Participants) | 6 | 6 | 12
    Stanford | 10.8 (2.4) | 9.7 (1.4) | 10.25 (2.3)
    BDC-UColorado: number analyzed (Participants) | 6 | 6 | 12
    BDC-UColorado | 9.2 (1.6) | 8.8 (0.4) | 9 (1.1)
    UVA: number analyzed (Participants) | 12 | 12 | 24
    UVA | 15.0 (1.4) | 14.8 (1.8) | 14.9 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 48 participated and completed the study (24 in UVA, 12 in Colorado, and 12 at Stanford). One subject signed consent but didn't met eligibility (no history of pump use), and five subjects left the study after a change in the Stanford camp dates (blizzard cancellation).
  Participants
    Stanford: number analyzed (Participants) | 6 | 6 | 12
    Stanford: Female | 3 | 3 | 6
    Stanford: Male | 3 | 3 | 6
    BDC-UColorado: number analyzed (Participants) | 6 | 6 | 12
    BDC-UColorado: Female | 3 | 3 | 6
    BDC-UColorado: Male | 3 | 3 | 6
    UVA: number analyzed (Participants) | 12 | 12 | 24
    UVA: Female | 6 | 4 | 10
    UVA: Male | 6 | 8 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 24 | 23 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Site [Count of Participants; unit: Participants]
  CA | 6 | 6 | 12
  CO | 6 | 6 | 12
  VA | 12 | 12 | 24
Height [Mean (Standard Deviation); unit: cm] — Population: 48 participated and completed the study (24 in UVA, 12 in Colorado, and 12 at Stanford). One subject signed consent but didn't met eligibility (no history of pump use), and five subjects left the study after a change in the Stanford camp dates (blizzard cancellation).
  cm
    Stanford: number analyzed (Participants) | 6 | 6 | 12
    Stanford | 143.9 (12) | 138.4 (13.4) | 141.15 (14.0)
    BDC-UColorado: number analyzed (Participants) | 6 | 6 | 12
    BDC-UColorado | 137.9 (8.9) | 136.5 (2.4) | 137.2 (6.3)
    UVA: number analyzed (Participants) | 12 | 12 | 24
    UVA | 166.6 (10.2) | 168.9 (8.7) | 167.8 (9.3)
Weight [Mean (Standard Deviation); unit: kg] — Population: 48 participated and completed the study (24 in UVA, 12 in Colorado, and 12 at Stanford). One subject signed consent but didn't met eligibility (no history of pump use), and five subjects left the study after a change in the Stanford camp dates (blizzard cancellation).
  kg
    Stanford: number analyzed (Participants) | 6 | 6 | 12
    Stanford | 41.2 (9.2) | 36.7 (4.4) | 38.9 (10.3)
    BDC-UColorado: number analyzed (Participants) | 6 | 6 | 12
    BDC-UColorado | 36.5 (10.7) | 31 (3.1) | 33.7 (8.0)
    UVA: number analyzed (Participants) | 12 | 12 | 24
    UVA | 60.1 (10.9) | 73.6 (16.8) | 66.9 (15.5)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: 48 participated and completed the study (24 in UVA, 12 in Colorado, and 12 at Stanford). One subject signed consent but didn't met eligibility (no history of pump use), and five subjects left the study after a change in the Stanford camp dates (blizzard cancellation).
  kg/m^2
    Stanford: number analyzed (Participants) | 6 | 6 | 12
    Stanford | 19.6 (1.5) | 18.9 (0.8) | 19.2 (3.3)
    BDC-UColorado: number analyzed (Participants) | 6 | 6 | 12
    BDC-UColorado | 18.9 (3.8) | 16.6 (1.6) | 17.8 (3.0)
    UVA: number analyzed (Participants) | 12 | 12 | 24
    UVA | 21.5 (2.4) | 25.7 (4.7) | 23.6 (4.2)
Diabetes Duration [Mean (Standard Deviation); unit: years] — Population: 48 participated and completed the study (24 in UVA, 12 in Colorado, and 12 at Stanford). One subject signed consent but didn't met eligibility (no history of pump use), and five subjects left the study after a change in the Stanford camp dates (blizzard cancellation).
  years
    Stanford: number analyzed (Participants) | 6 | 6 | 12
    Stanford | 4.7 (0.2) | 4.0 (0.7) | 4.3 (1.6)
    BDC-UColorado: number analyzed (Participants) | 6 | 6 | 12
    BDC-UColorado | 4.7 (2.8) | 4.8 (1.6) | 4.75 (2.2)
    UVA: number analyzed (Participants) | 12 | 12 | 24
    UVA | 6.7 (3.2) | 5.6 (2.4) | 6.1 (2.8)
Pump use [Mean (Standard Deviation); unit: years] — Population: 48 participated and completed the study (24 in UVA, 12 in Colorado, and 12 at Stanford). One subject signed consent but didn't met eligibility (no history of pump use), and five subjects left the study after a change in the Stanford camp dates (blizzard cancellation).
  years
    Stanford: number analyzed (Participants) | 6 | 6 | 12
    Stanford | 4.2 (1.7) | 3.3 (0.7) | 3.75 (1.7)
    BDC-UColorado: number analyzed (Participants) | 6 | 6 | 12
    BDC-UColorado | 4 (2.3) | 3.7 (2) | 3.8 (2.0)
    UVA: number analyzed (Participants) | 12 | 12 | 24
    UVA | 6.5 (3.5) | 4.9 (2.1) | 5.7 (2.9)
Daily Insulin Dose [Mean (Standard Deviation); unit: U/kg] — Population: 48 participated and completed the study (24 in UVA, 12 in Colorado, and 12 at Stanford). One subject signed consent but didn't met eligibility (no history of pump use), and five subjects left the study after a change in the Stanford camp dates (blizzard cancellation).
  U/kg
    Stanford: number analyzed (Participants) | 6 | 6 | 12
    Stanford | 0.8 (0.1) | 0.7 (0) | 0.7 (0.2)
    BDC-UColorado: number analyzed (Participants) | 6 | 6 | 12
    BDC-UColorado | 0.7 (0.3) | 0.7 (0.2) | 0.7 (0.2)
    UVA: number analyzed (Participants) | 12 | 12 | 24
    UVA | 0.8 (0.2) | 0.8 (0.2) | 0.8 (0.2)
Glycated hemoglobin [Mean (Standard Deviation); unit: %] — Population: 48 participated and completed the study (24 in UVA, 12 in Colorado, and 12 at Stanford). One subject signed consent but didn't met eligibility (no history of pump use), and five subjects left the study after a change in the Stanford camp dates (blizzard cancellation).
  %
    Stanford: number analyzed (Participants) | 6 | 6 | 12
    Stanford | 7.4 (0.7) | 7.2 (0.3) | 7.3 (0.6)
    BDC-UColorado: number analyzed (Participants) | 6 | 6 | 12
    BDC-UColorado | 7.3 (0.8) | 7.6 (0.7) | 7.4 (0.7)
    UVA: number analyzed (Participants) | 12 | 12 | 24
    UVA | 8.3 (1.5) | 8.0 (1.1) | 8.2 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Percent Time Spent Between 70 and 180 mg/dL
Description: The primary outcome was the percent time spent between 70 and 180 mg/dL during the 48hr study admission.
Time Frame: Overall [48hr study admission]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens." Data for three participants were excluded. For one subject, a software error resulted in prolonged AP system downtime. For a second subject, repeated pump occlusions resulted in prolonged system downtime. For the third subject, the Tandem pump was initialized with a sibling's pump settings resulting in strongly biased results.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 66.4 (16.4) | 53.9 (24.8)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 59.9 (19.5) | 57.7 (23.1)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 73.5 (8.4) | 50 (26.8)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.010, ANOVA — Primary statistical analysis between treatment groups was performed using univariate ANOVA with the treatment mode as a fixed factor. P value <0.05 was considered significant
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.089, ANOVA — Primary statistical analysis between treatment groups was performed using univariate ANOVA with age group as a fixed factor. P value <0.05 was considered significant
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.024, ANOVA — Primary statistical analysis between treatment groups was performed using univariate ANOVA with the treatment mode and age group as fixed factors. P value <0.05 was considered significant

2. Primary Outcome: Percent Time Spent Between 70 and 180 mg/dL
Description: This outcome looks at the percentage of time spent between 70 and 180 mg/dL during the Daytime, defined as 7am-11pm.
Time Frame: Daytime [7am - 11pm]
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 62.4 (18.8) | 54.8 (24.9)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 56.4 (22.7) | 59.6 (22.3)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 68.9 (11.1) | 50 (27.3)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.095, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.104, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.042, ANOVA — [p-value comment as in outcome 1, analysis 3]

3. Primary Outcome: Percent Time Spent Between 70 and 180 mg/dL
Description: This outcome looks at the percentage of time spent between 70 and 180 mg/dL during the Overnight, defined as 11pm-7am.
Time Frame: Overnight [11pm - 7am]
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 78.6 (20.3) | 50.9 (34.2)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 70.6 (24) | 52 (34.3)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 87.3 (10.8) | 49.9 (35.6)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.065, ANOVA — [p-value comment as in outcome 1, analysis 3]

4. Primary Outcome: Percent Time Spent Between 70 and 180 mg/dL
Description: This outcome looks at the percentage of time spent between 70 and 180 mg/dL during the Skiing periods, defined as 9:30am-noon and 1:30pm-4pm.
Time Frame: Skiing [9:30am-noon and 1:30pm-4pm]
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 57.8 (27.3) | 55.9 (31.1)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 50 (30.7) | 65.2 (24)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 66.4 (21.1) | 46.6 (35.5)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.063, ANOVA — [p-value comment as in outcome 1, analysis 3]

5. Secondary Outcome: Percent Time Spent <50 mg/dL
Description: The percentage of time spent below 50 mg/dL during the Overall period. CGM measured blood sugar values below 50 mg/dL falls into the range of hypoglycemia which have the potential to lead to unconsciousness or death. Thus, less time below 50 mg/dL is considered a better outcome.
Time Frame: Overall [48hr study admission]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 0 [0 to 0] | 0 [0 to 0]
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 0 [0 to 0] | 0 [0 to 0.1]
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — Primary statistical analysis between treatment groups was performed using Wilcoxon signed-rank test with the treatment mode as a fixed factor. P value <0.05 was considered significant
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — Primary statistical analysis between treatment groups was performed using Wilcoxon signed-rank test with age group as a fixed factor. P value <0.05 was considered significant
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — Primary statistical analysis between treatment groups was performed using Wilcoxon signed-rank test with the treatment mode and age group as fixed factors. P value <0.05 was considered significant

6. Secondary Outcome: Percent Time Spent <54 mg/dL
Description: The percentage of time spent below 54 mg/dL during the Overall period. CGM measured blood sugar values below 54 mg/dL falls into the range of hypoglycemia which have the potential to lead to unconsciousness or death. Thus, less time below 54 mg/dL is considered a better outcome.
Time Frame: Overall [48hr study admission]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 0 [0 to 0] | 0 [0 to 0.1]
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 0 [0 to 0] | 0 [0 to 0.5]
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 0 [0 to 0.2] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 3]

7. Secondary Outcome: Percent Time Spent <60 mg/dL
Description: The percentage of time spent below 60 mg/dL during the Overall period. CGM measured blood sugar values below 60 mg/dL falls into the range of hypoglycemia which have the potential to lead to unconsciousness or death. Thus, less time below 60 mg/dL is considered a better outcome.
Time Frame: Overall [48hr study admission]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 0 [0 to 0.8] | 0 [0 to 0.6]
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 0 [0 to 0.3] | 0 [0 to 0.9]
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 0.5 [0 to 1.6] | 0 [0 to 0.5]
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 3]

8. Secondary Outcome: Percent Time Spent <70 mg/dL
Description: The percentage of time spent below 70 mg/dL during the Overall period. CGM measured blood sugar values below 70 mg/dL falls into the range of hypoglycemia which have the potential to lead to unconsciousness or death. Thus, less time below 70 mg/dL is considered a better outcome.
Time Frame: Overall [48hr study admission]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 2 [0.5 to 3.8] | 0.8 [0 to 3.7]
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 0.8 [0 to 1.6] | 0.8 [0.4 to 3]
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 3.3 [2.3 to 4.5] | 0.9 [0 to 4.5]
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.062, ANOVA — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 5, analysis 3]

9. Secondary Outcome: Percent Time Spent >180 mg/dL
Description: The percentage of time spent above 180 mg/dL during the overall period. CGM measured blood sugar values above 180 mg/dL are considered to be undesirable. Thus, less time spent above 180 mg/dL is considered a positive outcome.
Time Frame: Overall [48hr study admission]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 31.4 (17.6) | 43 (24.5)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 39 (20.5) | 40.5 (23.1)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 22.9 (8.2) | 45.5 (26.7)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.015, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.199, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.025, ANOVA — [p-value comment as in outcome 1, analysis 3]

10. Secondary Outcome: Percent Time Spent >250 mg/dL
Description: The percentage of time spent above 250 mg/dL during the Overall period. CGM measured blood sugar values above 250 mg/dL are considered to be undesirable. Thus, less time spent above 250 mg/dL is considered a positive outcome.
Time Frame: Overall [48hr study admission]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 10.4 (11.4) | 16 (13.6)
  School-age [6 -12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6 -12 years old] | 14.8 (14) | 13.2 (12.5)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 5.6 (4.9) | 18.8 (14.5)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.059, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.064, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.017, ANOVA — [p-value comment as in outcome 1, analysis 3]

11. Secondary Outcome: Percent Time Spent >300 mg/dL
Description: The percentage of time spent above 300 mg/dL. CGM measured blood sugar values above 300 mg/dL are considered to be undesirable. Thus, less time spent above 300 mg/dL is considered a positive outcome.
Time Frame: Overall [48hr study admission]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 3.9 (5.9) | 6.9 (6.7)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 6.5 (7.2) | 6.6 (6.6)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 1 (1.3) | 7.3 (7)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.034, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.074, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.034, ANOVA — [p-value comment as in outcome 1, analysis 3]

12. Secondary Outcome: Mean Glucose
Description: Mean glucose is a measure of the average CGM value in mg/dL during the Overall period. A lower value, without approaching hypoglycemia, is indicative of a desirable outcome.
Time Frame: Overall [48hr study admission]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
mg/dL
  All | 161 (29.9) | 176.8 (36.5)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 175.9 (33.9) | 174.5 (30.7)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 144.5 (11.7) | 179 (42.7)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.023, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.016, ANOVA — [p-value comment as in outcome 1, analysis 3]

13. Secondary Outcome: Glucose Variability
Description: Variability of glucose during the Overall period
Time Frame: Overall [48hr study admission]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: coefficient of variation
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
coefficient of variation
  All | 34.2 (6.1) | 33.9 (8.4)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 32.4 (5.3) | 33.2 (8)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 36.2 (6.6) | 34.6 (9)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 3]

14. Secondary Outcome: Insulin
Description: Amount (U/kg) of insulin administered during the Overall period
Time Frame: Overall [48hr study admission]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
U/kg
  All | 40.5 (16.7) | 43.9 (28.4)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 29.5 (10.9) | 21.4 (8.4)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 52.7 (13.1) | 66.3 (22.8)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.081, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 3]

15. Secondary Outcome: Carbohydrate (CHO) Treatment
Description: The amount of carbohydrates in grams administered as treatment for hypoglycemia in the Overall period.
Time Frame: Overall [48hr study admission]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
grams
  All | 45.5 (27.8) | 57.7 (57.8)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 42.1 (27.3) | 55.8 (36.1)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 49.3 (29.2) | 59.6 (75.4)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 3]

16. Secondary Outcome: Percent Time Spent <50 mg/dL
Description: The percentage of time spent below 50 mg/dL during the Daytime period. CGM measured blood sugar values below 50 mg/dL falls into the range of hypoglycemia which have the potential to lead to unconsciousness or death. Thus, less time below 50 mg/dL is considered a better outcome.
Time Frame: Daytime [7am - 11pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 0 [0 to 0] | 0 [0 to 0]
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 0 [0 to 0] | 0 [0 to 0]
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 3]

17. Secondary Outcome: Percent Time Spent <54 mg/dL
Description: The percentage of time spent below 54 mg/dL during the Daytime period. CGM measured blood sugar values below 54 mg/dL falls into the range of hypoglycemia which have the potential to lead to unconsciousness or death. Thus, less time below 54 mg/dL is considered a better outcome.
Time Frame: Daytime [7am - 11pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 0 [0 to 0] | 0 [0 to 0]
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 0 [0 to 0] | 0 [0 to 0.1]
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 3]

18. Secondary Outcome: Percent Time Spent <60 mg/dL
Description: The percentage of time spent below 60 mg/dL during the Daytime period. CGM measured blood sugar values below 60 mg/dL falls into the range of hypoglycemia which have the potential to lead to unconsciousness or death. Thus, less time below 60 mg/dL is considered a better outcome.
Time Frame: Daytime [7am - 11pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 0 [0 to 0.3] | 0 [0 to 0.1]
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 0 [0 to 0] | 0 [0 to 0.8]
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 0 [0 to 0.8] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 3]

19. Secondary Outcome: Percent Time Spent <70 mg/dL
Description: The percentage of time spent below 70 mg/dL during the Daytime period. CGM measured blood sugar values below 70 mg/dL falls into the range of hypoglycemia which have the potential to lead to unconsciousness or death. Thus, less time below 70 mg/dL is considered a better outcome.
Time Frame: Daytime [7am - 11pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 1 [0 to 3.3] | 0.8 [0 to 2]
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 0.7 [0 to 1.7] | 1 [0.5 to 2.7]
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 2.5 [0.4 to 4.7] | 0.7 [0 to 1.8]
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 3]

20. Secondary Outcome: Percent Time Spent >180 mg/dL
Description: The percentage of time spent above 180 mg/dL during the Daytime period. CGM measured blood sugar values above 180 mg/dL are considered to be undesirable. Thus, less time spent above 180 mg/dL is considered a positive outcome.
Time Frame: Daytime [7am - 11pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 35.7 (19.8) | 42.5 (24.9)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 42.6 (23.7) | 38.4 (22.4)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 28.1 (11.3) | 46.5 (27.6)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.124, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.187, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.040, ANOVA — [p-value comment as in outcome 1, analysis 3]

21. Secondary Outcome: Percent Time Spent >250 mg/dL
Description: The percentage of time spent above 250 mg/dL during the Daytime period. CGM measured blood sugar values above 250 mg/dL are considered to be undesirable. Thus, less time spent above 250 mg/dL is considered a positive outcome.
Time Frame: Daytime [7am - 11pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 12.1 (13.6) | 16.9 (14.4)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 17.1 (16.3) | 13.3 (12)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 6.6 (6.9) | 20.4 (16.3)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.108, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.053, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.010, ANOVA — [p-value comment as in outcome 1, analysis 3]

22. Secondary Outcome: Percent Time Spent >300 mg/dL
Description: The percentage of time spent above 300 mg/dL during the Daytime period. CGM measured blood sugar values above 300 mg/dL are considered to be undesirable. Thus, less time spent above 300 mg/dL is considered a positive outcome.
Time Frame: Daytime [7am - 11pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 4.6 (7.2) | 7.3 (7.5)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 7.6 (9) | 6.5 (6.4)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 1.3 (1.7) | 8.1 (8.7)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.080, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.038, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.016, ANOVA — [p-value comment as in outcome 1, analysis 3]

23. Secondary Outcome: Mean Glucose
Description: Mean glucose is a measure of the average CGM value in mg/dL during the Daytime period. A lower value, without approaching hypoglycemia, is indicative of a desirable outcome.
Time Frame: Daytime [7am - 11pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
mg/dL
  All | 166.9 (34) | 177.2 (37.6)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 180.3 (40.6) | 170.4 (30.1)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 152 (16.4) | 183.9 (44.1)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.111, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.130, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.017, ANOVA — [p-value comment as in outcome 1, analysis 3]

24. Secondary Outcome: Glucose Variability
Description: Variability of glucose during the Daytime period
Time Frame: Daytime [7am - 11pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: coefficient of variation
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
coefficient of variation
  All | 33.5 (4.8) | 34.2 (8.2)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 32.2 (3.3) | 35.3 (8.1)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 34.9 (5.9) | 33.2 (8.5)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 3]

25. Secondary Outcome: Insulin
Description: Amount (U/kg) of insulin administered during the Daytime period
Time Frame: Daytime [7am - 11pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
U/kg
  All | 30.9 (13.1) | 32.7 (20.4)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 22.1 (8) | 16.3 (6.2)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 40.7 (10.5) | 49 (15.8)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.044, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 3]

26. Secondary Outcome: CHO Treatment
Description: The amount of carbohydrates in grams administered as treatment for hypoglycemia in the Daytime period.
Time Frame: Daytime [7am - 11pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
grams
  All | 38.5 (25.2) | 47.5 (50.2)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 35.1 (23.6) | 46.8 (29.1)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 42.3 (27.6) | 48.2 (66.5)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 3]

27. Secondary Outcome: Percent Time Spent <50 mg/dL
Description: The percentage of time spent below 50 mg/dL during the Overnight period. CGM measured blood sugar values below 50 mg/dL falls into the range of hypoglycemia which have the potential to lead to unconsciousness or death. Thus, less time below 50 mg/dL is considered a better outcome.
Time Frame: Overnight [11pm - 7am]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 0 [0 to 0] | 0 [0 to 0]
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 0 [0 to 0] | 0 [0 to 0]
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 3]

28. Secondary Outcome: Percent Time Spent <54 mg/dL
Description: The percentage of time spent below 54 mg/dL during the Overnight period. CGM measured blood sugar values below 54 mg/dL falls into the range of hypoglycemia which have the potential to lead to unconsciousness or death. Thus, less time below 54 mg/dL is considered a better outcome.
Time Frame: Overnight [11pm - 7am]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 0 [0 to 0] | 0 [0 to 0]
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 0 [0 to 0] | 0 [0 to 0]
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 3]

29. Secondary Outcome: Percent Time Spent <60 mg/dL
Description: The percentage of time spent below 60 mg/dL during the Overnight period. CGM measured blood sugar values below 60 mg/dL falls into the range of hypoglycemia which have the potential to lead to unconsciousness or death. Thus, less time below 60 mg/dL is considered a better outcome.
Time Frame: Overnight [11pm - 7am]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 0 [0 to 1] | 0 [0 to 0]
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 0 [0 to 0] | 0 [0 to 0]
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 0.5 [0 to 1.8] | 0 [0 to 0.5]
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.141, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.149, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 3]

30. Secondary Outcome: Percent Time Spent <70 mg/dL
Description: as for outcome 8
Time Frame: Overnight [11pm - 7am]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 0 [0 to 8.2] | 0 [0 to 6.4]
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 0 [0 to 0] | 0 [0 to 0]
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 6.1 [0.3 to 9.7] | 0 [0 to 8.2]
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.094, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 3]

31. Secondary Outcome: Percent Time Spent Between 70 and 150 mg/dL
Description: This outcome looks at the percentage of time spent between 70 and 150 mg/dL during the Overnight, defined as 11pm-7am.
Time Frame: Overnight [11pm - 7am]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 60.8 (26.5) | 32.1 (33.2)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 45.5 (27.7) | 24.7 (28.5)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 77.6 (10.4) | 39.5 (37.1)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p < 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.033, ANOVA — [p-value comment as in outcome 1, analysis 3]

32. Secondary Outcome: Percent Time Spent >180 mg/dL
Description: The percentage of time spent above 180 mg/dL during the Overnight period. CGM measured blood sugar values above 180 mg/dL are considered to be undesirable. Thus, less time spent above 180 mg/dL is considered a positive outcome.
Time Frame: Overnight [11pm - 7am]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 18.2 (21.4) | 44.5 (37)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 28.2 (23.3) | 46.7 (34.1)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 7.1 (12.5) | 42.3 (41.1)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.001, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.111, ANOVA — [p-value comment as in outcome 1, analysis 3]

33. Secondary Outcome: Percent Time Spent >250 mg/dL
Description: The percentage of time spent above 250 mg/dL during the Overnight period. CGM measured blood sugar values above 250 mg/dL are considered to be undesirable. Thus, less time spent above 250 mg/dL is considered a positive outcome.
Time Frame: Overnight [11pm - 7am]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 5.3 (13.5) | 13.2 (19)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 7.7 (17) | 12.7 (20.2)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 2.7 (8.4) | 13.7 (18.6)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.118, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 3]

34. Secondary Outcome: Percent Time Spent >300 mg/dL
Description: The percentage of time spent above 300 mg/dL during the Overnight period. CGM measured blood sugar values above 300 mg/dL are considered to be undesirable. Thus, less time spent above 300 mg/dL is considered a positive outcome.
Time Frame: Overnight [11pm - 7am]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 1.8 (7.8) | 5.8 (9.5)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 3.2 (10.8) | 6.7 (11.7)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 0.2 (0.6) | 4.8 (7)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.116, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 3]

35. Secondary Outcome: Mean Glucose
Description: Mean glucose is a measure of the average CGM value in mg/dL during the Overnight period. A lower value, without approaching hypoglycemia, is indicative of a desirable outcome.
Time Frame: Overnight [11pm - 7am]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
mg/dL
  All | 142.9 (36) | 175.4 (52.7)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 162.4 (37) | 187.1 (39.9)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 121.6 (19.7) | 163.8 (62.6)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.005, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.193, ANOVA — [p-value comment as in outcome 1, analysis 3]

36. Secondary Outcome: Glucose Variability
Description: Variability of glucose during the Overnight period
Time Frame: Overnight [11pm - 7am]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: coefficient of variation
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
coefficient of variation
  All | 24.5 (9.9) | 24.3 (11.6)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 22.6 (8.9) | 21 (13.3)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 26.5 (10.9) | 27.6 (9)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.106, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 3]

37. Secondary Outcome: Insulin
Description: Amount (U/kg) of insulin administered during the Overnight period
Time Frame: Overnight [11pm - 7am]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
U/kg
  All | 7.5 (3.1) | 9.4 (10)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 6.1 (3) | 4.1 (2.5)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 9 (2.6) | 14.8 (11.9)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.157, ANOVA — [p-value comment as in outcome 1, analysis 3]

38. Secondary Outcome: CHO Treatment
Description: The amount of carbohydrates in grams administered as treatment for hypoglycemia in the Overnight period.
Time Frame: Overnight [11pm - 7am]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
grams
  All | 2.8 (8.3) | 5.5 (12.4)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 3.4 (10) | 4 (9.7)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 2.1 (6.5) | 7 (14.9)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 3]

39. Secondary Outcome: Percent Time Spent <50 mg/dL
Description: The percentage of time spent below 50 mg/dL during the Skiing period. CGM measured blood sugar values below 50 mg/dL falls into the range of hypoglycemia which have the potential to lead to unconsciousness or death. Thus, less time below 50 mg/dL is considered a better outcome.
Time Frame: Skiing [9:30am-noon and 1:30pm-4pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 0 [0 to 0] | 0 [0 to 0]
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 0 [0 to 0] | 0 [0 to 0]
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 3]

40. Secondary Outcome: Percent Time Spent <54 mg/dL
Description: The percentage of time spent below 54 mg/dL during the Skiing period. CGM measured blood sugar values below 54 mg/dL falls into the range of hypoglycemia which have the potential to lead to unconsciousness or death. Thus, less time below 54 mg/dL is considered a better outcome.
Time Frame: Skiing [9:30am-noon and 1:30pm-4pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 0 [0 to 0] | 0 [0 to 0]
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 0 [0 to 0] | 0 [0 to 0]
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 3]

41. Secondary Outcome: Percent Time Spent <60 mg/dL
Description: The percentage of time spent below 60 mg/dL during the Skiing period. CGM measured blood sugar values below 60 mg/dL falls into the range of hypoglycemia which have the potential to lead to unconsciousness or death. Thus, less time below 60 mg/dL is considered a better outcome.
Time Frame: Skiing [9:30am-noon and 1:30pm-4pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 0 [0 to 0] | 0 [0 to 0]
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 0 [0 to 0] | 0 [0 to 0]
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 3]

42. Secondary Outcome: Percent Time Spent <70 mg/dL
Description: The percentage of time spent below 70 mg/dL during the Skiing period. CGM measured blood sugar values below 70 mg/dL falls into the range of hypoglycemia which have the potential to lead to unconsciousness or death. Thus, less time below 70 mg/dL is considered a better outcome.
Time Frame: Skiing [9:30am-noon and 1:30pm-4pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 0 [0 to 0.8] | 0 [0 to 0.4]
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 0 [0 to 0.8] | 0 [0 to 1.9]
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 0 [0 to 0.8] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 5, analysis 3]

43. Secondary Outcome: Percent Time Spent >180 mg/dL
Description: The percentage of time spent above 180 mg/dL during the Skiing period. CGM measured blood sugar values above 180 mg/dL are considered to be undesirable. Thus, less time spent above 180 mg/dL is considered a positive outcome.
Time Frame: Skiing [9:30am-noon and 1:30pm-4pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 41.4 (27.8) | 41.5 (30.3)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 49.3 (31.4) | 33.4 (23.4)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 32.8 (21.5) | 49.5 (35)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.073, ANOVA — [p-value comment as in outcome 1, analysis 3]

44. Secondary Outcome: Percent Time Spent >250 mg/dL
Description: The percentage of time spent above 250 mg/dL during the Skiing period. CGM measured blood sugar values above 250 mg/dL are considered to be undesirable. Thus, less time spent above 250 mg/dL is considered a positive outcome.
Time Frame: Skiing [9:30am-noon and 1:30pm-4pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 14.4 (17.3) | 18.2 (20.4)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 19.8 (20.7) | 14.4 (16.4)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 8.5 (10.6) | 22 (23.8)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.064, ANOVA — [p-value comment as in outcome 1, analysis 3]

45. Secondary Outcome: Percent Time Spent >300 mg/dL
Description: The percentage of time spent above 300 mg/dL during the Skiing period. CGM measured blood sugar values above 300 mg/dL are considered to be undesirable. Thus, less time spent above 300 mg/dL is considered a positive outcome.
Time Frame: Skiing [9:30am-noon and 1:30pm-4pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
percentage of time
  All | 5.9 (11.1) | 7.5 (10.9)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 9.2 (14.6) | 8.1 (10.5)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 2.3 (3.2) | 6.9 (11.7)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 3]

46. Secondary Outcome: Mean Glucose
Description: Mean glucose is a measure of the average CGM value in mg/dL during the Skiing period. A lower value, without approaching hypoglycemia, is indicative of a desirable outcome.
Time Frame: Skiing [9:30am-noon and 1:30pm-4pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
mg/dL
  All | 173.2 (44.7) | 178 (47.4)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 185.3 (53.8) | 167.5 (33.3)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 159.8 (29) | 188.5 (57.8)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.104, ANOVA — [p-value comment as in outcome 1, analysis 3]

47. Secondary Outcome: Glucose Variability
Description: Variability of glucose during the Skiing period
Time Frame: Skiing [9:30am-noon and 1:30pm-4pm
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: coefficient of variation
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
coefficient of variation
  All | 30.2 (7.7) | 29.9 (10.5)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 30 (9.3) | 35.2 (10.2)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 30.3 (6) | 24.5 (7.9)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.198, ANOVA — [p-value comment as in outcome 1, analysis 3]

48. Secondary Outcome: Insulin
Description: Amount (U/kg) of insulin administered during the Skiing period
Time Frame: Skiing [9:30am-noon and 1:30pm-4pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
U/kg
  All | 6.8 (2.6) | 6.6 (5.8)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 6.6 (2.4) | 5 (3.1)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 6.9 (2.9) | 8.1 (7.4)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.105, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p = 0.001, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 3]

49. Secondary Outcome: CHO Treatment
Description: The amount of carbohydrates in grams administered as treatment for hypoglycemia in the Skiing period.
Time Frame: Skiing [9:30am-noon and 1:30pm-4pm]
Population: The "All" row is the combined total of participants in the following rows "School-age" and "Teens."
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Experimental AP Group | Control SAP Group
Number analyzed (Participants) | 21 | 24
grams
  All | 13.4 (14.8) | 14.6 (19.3)
  School-age [6-12 years old]: number analyzed (Participants) | 11 | 12
  School-age [6-12 years old] | 10.1 (9) | 14.3 (14.7)
  Teens [13-18 years old]: number analyzed (Participants) | 10 | 12
  Teens [13-18 years old] | 17.1 (19.3) | 14.9 (23.7)
Statistical Analysis 1: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Experimental AP Group vs Control SAP Group; Test type: Other; p > 0.2, ANOVA — [p-value comment as in outcome 1, analysis 3]

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Control SAP Group | Experimental AP Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

LIMITATIONS AND CAVEATS:
Data for 3 participants were excluded. Subject 1: a software error resulted in prolonged AP system downline. The error was identified in data analysis; Subject 2: repeated pump occlusion resulted in prolonged system downtime; Subject 3: study pump initialized with siblings pump settings resulting in strong biased results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-01-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT03369067/Prot_SAP_002.pdf
  • Informed Consent Form (2018-01-03): https://cdn.clinicaltrials.gov/large-docs/67/NCT03369067/ICF_001.pdf